CLINICAL TRIAL: NCT05401799
Title: Efficacy of the Barrett Upper Extremity Robot (BURT) for Improving Upper Extremity Strength and Function During Inpatient Rehabilitation Following Stroke.
Brief Title: BURT Efficacy in Improving Upper Extremity Strength and Function During Post-stroke Inpatient Rehabilitation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sunnyview Rehabilitation Hospital (Other)
Collaborators: Gaylord Hospital (Unknown)
Responsible Party: Principal Investigator, Casey Cowan, Occupational Therapist, Sunnyview Rehabilitation Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 22-0324-1
Record Dates: First submitted 2022-05-10; First posted 2022-06-02 (Actual); Last update posted 2025-05-18 (Actual); Status verified 2025-05

CONDITIONS: Stroke; Stroke, Acute; Cerebral Vascular Accident; Cerebral Vascular Accident (CVA)/Stroke
Keywords: BURT; Upper extremity function; Inpatient rehabilitation; Upper extremity robotics
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Conventional Upper Extremity Neuroeducation (Active Comparator): 74 patients will receive the standard occupational therapy sessions that they would normally receive during their IRF stay. UE neuroeducation sessions are typically focused on improving strength and mobility of the upper arm. Clinicians will not be given instructions on how to run their sessions, however they will not be allowed to use BURT. Other devices that would normally be used during neuro-educational sessions (including X-cite, electrical stimulation and RT-300) will be allowed for use in this group. The therapists will track the activity, level of assistance and time provided in a tracking sheet, as well as document any adverse events that may occur
  Interventions: Procedure: Other Occupational Therapy
- BURT Upper Extremity (Experimental): As part of routine therapy, 74 patients will receive up to 5 sessions per week of BURT UE therapy in place of conventional neuro re-education. Patients in this arm of the study will receive any conventional therapy during the remainder of their treatment sessions. When using BURT, therapists will track the activity, level of assistance and time provided in a tracking sheet, as well as document any adverse events that may occur.
  Interventions: Device: BURT; Procedure: Other Occupational Therapy

INTERVENTIONS:
Device: BURT — Use of Barrett Upper extremity Robot (BURT) to improve strength and mobility of hemiplegic upper extremity.
  Arms: BURT Upper Extremity
Procedure: Other Occupational Therapy — Standard occupational therapy sessions will be 60-90 minutes a day and are UE neuroeducation sessions are typically focused on improving strength and mobility of the hemipelagic arm.

SUMMARY:
The Barrett Upper Extremity Robot (BURT) is an FDA-approved upper extremity robot that assists patients with both passive and active range of motion while providing adjustable resistance (Barrett_Medical. Robotic Assist Rehabilitation Made Easy. https://medical.barrett.com/). Activities are directed by therapists and encourage patient involvement through video game activities providing active proprioceptive, vibrational, visual and auditory feedback. Engaging and colorful games are beneficial in holding patients' interest, and gravity assistance may also allow for increased repetition in the face of patient fatigue.

In this prospective study, the investigators will determine if a standardized BURT Upper Extremity (UE) program can be consistently implemented within an acute inpatient rehabilitation facility (IRF). In addition, the investigators will see if patients who receive BURT have improved UE mobility and function as a result. The investigators will also study the perceived enjoyment and value of the intervention by patients, and perceived value by therapists.

Because BURT therapy is able to provide more repetitions of upper extremity movement in a shorter length of time than conventional therapy, the investigators hypothesize that patients who participate in neuro re-education activities using BURT will achieve greater improvements in strength, upper extremity function, fine motor coordination, activities of daily living and mobility during their time in an IRF than patients receiving conventional therapy.

In this study, eligible patients admitted to Sunnyview Rehabilitation Hospital (SRH) for rehabilitation following stroke will be randomized to receive conventional or BURT therapy. Meaningful clinical benchmarks for upper extremity function, tone, fine motor coordination, activities of daily living and mobility will be assessed using the Upper Extremity Motor Assessment Scale (UE-MAS)(Zelter, 2010), manual muscle testing (MMT), Modified Ashworth Scale (MAS) (Figueiredo, 2011) and the 9-hole peg test (9HPT)(Figueiredo, 2011). The investigators also hypothesize that patients in the BURT cohort will report greater value/usefulness and interest/enjoyment.

ELIGIBILITY:
Inclusion Criteria:

* Inpatient at Sunnyview Rehabilitation Hospital
* >/= 18 years
* Unilateral stroke
* UE paresis affected arm with 3-/5 or less manual muscle testing throughout

Exclusion Criteria:

>30 days post stroke

* Severe Neglect
* Bilateral stroke
* Prior stroke with residual deficits
* Patients receiving prism adaptation treatment
* Comorbid neurological disorders
* Upper limb comorbidities that could limit functional improvement (UE arthritis pain, UE fracture, fixed contracture not allowing for proper device alignment)
* Severe shoulder subluxation that cannot be accommodated by the device
* Severe osteoporosis
* Unable to follow simple directions
* Unable to tolerate sitting 30 minutes
* Expected length of stay (LOS) < 15 days.

Ages: 18 Years to 115 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2025-02-17 (Actual); Study Completion 2025-02-17 (Actual)

PRIMARY OUTCOMES:
UE Motor Assessment Scale (UE-MAS) | T2(Day 20-23) - T0 (Day 4-6)
  Used to assess motor functions in the affected upper extremity following a stroke. This evaluation uses task-oriented techniques instead of isolated movement patterns.
UE Motor Assessment Scale (UE-MAS) | T1 (Day 12-14) - T0 (Day 4-6)
  Used to assess motor functions in the affected upper extremity following a stroke. This evaluation uses task-oriented techniques instead of isolated movement patterns.
Manual Muscle Testing (MMT) | T2(Day 20-23) - T0 (Day 4-6)
  Used to assess the strength in a persons upper extremity based on various planes of movement. This is the most commonly used strength assessment.
Manual Muscle Testing (MMT) | T1 (Day 12-14) - T0 (Day 4-6)
  Used to assess the strength in a persons upper extremity based on various planes of movement. This is the most commonly used strength assessment.
Modified Ashworth Scale (MAS) | T2(Day 20-23) - T0 (Day 4-6)
  The modified Ashworth Scale is the primary measure for muscle spasticity in the upper extremities for patients with neurological conditions.
Modified Ashworth Scale (MAS) | T1 (Day 12-14) - T0 (Day 4-6)
  The modified Ashworth Scale is the primary measure for muscle spasticity in the upper extremities for patients with neurological conditions.
9 Hole Peg Test (9HPT) | T2(Day 20-23) - T0 (Day 4-6)
  The 9HPT is a standardized test that measures manual dexterity.
9 Hole Peg Test (9HPT) | T1 (Day 12-14) - T0 (Day 4-6)
  The 9HPT is a standardized test that measures manual dexterity.

SECONDARY OUTCOMES:
GG Scores for Self-Care Items | Change from admission to discharge, up to 55 days
  standardized assessments of functional independence for feeding, bathing, toileting, footwear, upper and lower body dressing and oral hygiene.
GG Scores for Mobility items | Change from admission to discharge, up to 55 days
  standardized assessments of functional independence for bed mobility and transfers.

CONTACTS AND LOCATIONS:
Overall Officials: Casey Cowan, MS OTR/L, Principal Investigator — Sunnyview Rehabilitation Hospital; Emily Steenburgh, MS OTR/L, Principal Investigator — Sunnyview Rehabilitation Hospital
Locations (2):
- United States (2):
  - Gaylord Hospital, Wallingford, Connecticut
  - Sunnyview Rehabilitation Hospital, Schenectady, New York

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Barrett_Medical. Robotic Assist Rehabilitation Made Easy. https://medical.barrett.com/
- [Background] Zelter L. 2010. Motor Assessment Scale (MAS). https://strokengine.ca/en/assessments/motor-assessment-scale-mas/#:~:text=The%20Motor%20Assessment%20Scale%20(MAS,leakage%20from%20a%20blood%20vessel.
- [Background] Figueiredo S ZL. 2011. Modified Ashworth Scale. https://strokengine.ca/en/assessments/modified-ashworth-scale/
- [Background] Figueiredo S. 2011. Nine Hole Peg Test (NHPT). https://strokengine.ca/en/assessments/nine-hole-peg-test-nhpt/